CLINICAL TRIAL: NCT05652816
Title: Substitute Graft for Burns Using Biological Graft Seeded With Autologous Keratinocyte Co-cultured With Stem Cells
Brief Title: Biological Skin Graft With Keratinocyte-stem Cell Co-cultre for Burn Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Aditya Wardhana, Head of Burns Unit, Cipto Mangunkusumo National Hospital, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KET-866/ETIK/2021
Record Dates: First submitted 2022-11-29; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Burn Degree Second; Burn Degree Third
Keywords: artificial skin graft; keratinocyte; amnion epithelial stem cells; burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STSG (Split-Thickness Skin Graft) (Sham Comparator): Patients treated with the standard treatment; autologous skin graft
  Interventions: Procedure: Split-thickness skin graft
- Amnion Bilayer Only (Experimental): Patients treated with artificial graft only
  Interventions: Biological: Artificial skin graft
- Amnion Bilayer seeded with co-culture (Experimental): Patients treated with artificial graft seeded with autologous keratinocyte co-cultured with amnion epithelial stem cells
  Interventions: Biological: Artificial skin graft co-culture

INTERVENTIONS:
Procedure: Split-thickness skin graft — Transplantation of autologous skin to burn area
  Arms: STSG (Split-Thickness Skin Graft)
Biological: Artificial skin graft — Decellularized amnion membrane formed into 3-D matrix
  Arms: Amnion Bilayer Only
Biological: Artificial skin graft co-culture — Decellularized amnion membrane formed into 3-D matrix seeded with autologous keratinocyte co-cultured with amnion epithelial stem cells
  Arms: Amnion Bilayer seeded with co-culture

SUMMARY:
The goal of this clinical trial is to test whether artificial skin graft can substitute autologous skin graft in current burn treatment. The main question it aims to answer is:

• Can artificial skin graft result in better wound healing compared to the current burn treatment; autologous skin graft?

You will:

* Undergo debridement surgery
* Receive artificial skin graft as an alternative to autologous skin graft
* Undergo biopsy procedure of burn area

If there is a comparison group: Researchers will compare autologous skin graft group to see the wound healing process

DETAILED DESCRIPTION:
Burn caused by working accidents occurs mostly in the male population of productive age (68.68%). Up to this date, the only treatment for grade 2B-3 burns patients in Indonesia is skin transplantation taken from their own body (autologous skin graft). This treatment has several drawbacks in which repeated surgery is sometimes necessary, the source of skin in patients with wide area of burn is limited, and patients that are in the elder age and have comorbidities have high mortality risk.

In order to find an alternative for autologous skin graft therapy, a combination of tissue engineering and stem cell therapy is used to invent an artificial skin graft. The present study attempts to evaluate the efficacy of artificial skin graft seeded with autologous keratinocyte and stem cells towards wound healing in burn patients. The artificial graft used in this study is amnion bilayer; a graft that was decellularized to remove donor's cells and then layered to form into 3-D.

To evaluate the efficacy, biopsies are taken from the burn area of patients to evaluate the histoarchitecture of patients' tissue by histological staining (H&E and Movat's pentachrome, IHC collagen I, collagen III, vWF, and alpha-SMA) and measure the relative gene expression by qPCR. For clinical data, burn area calculation using Rule of 9 method and thermography measurement using FLIRONE. Furthermore, systemic evaluation of patients are done by monitoring the procalcitonin, lactate, mean arterial pressure, gradation of wound, and sensory of burn area. The evaluation and measurement mentioned above are then compared to patients treated with the current available therapy; autologous skin graft. The artificial skin graft is hoped to result in equal, if not better, wound healing in burn patients compared to autologous skin graft. The investigators hope that artificial skin graft can be an option, other than autologous skin graft, in treating burn patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 55
* Area of burn <50%
* Acute phase burn (<120 hrs)
* Have not undergo any surgery for burn treatment

Exclusion Criteria:

* Immunocompromised
* Have comorbidities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Burn thickness | Day of surgery
  Thickness of burn evaluation using Rule of 9
Burn thickness | Day 7 after surgery
  Thickness of burn evaluation using Rule of 9
Burn thickness | Day 14 after surgery
  Thickness of burn evaluation using Rule of 9
Burn thermography | Day of surgery
  Thermography evaluation using FLIRONE
Burn thermography | Day 7 after surgery
  Thermography evaluation using FLIRONE
Burn thermography | Day 14 after surgery
  Thermography evaluation using FLIRONE
Systemic clinical evaluation | Day of surgery
  Mean arterial pressure measurement
Systemic clinical evaluation | Day 7 after surgery
  Mean arterial pressure measurement
Systemic clinical evaluation | Day 14 after surgery
  Mean arterial pressure measurement
Systemic clinical evaluation | Day of surgery
  lactate measurement
Systemic clinical evaluation | Day 7 after surgery
  lactate measurement
Systemic clinical evaluation | Day 14 after surgery
  lactate measurement
Systemic clinical evaluation | Day of surgery
  procalcitonin measurement
Systemic clinical evaluation | Day 7 after surgery
  procalcitonin measurement
Systemic clinical evaluation | Day 14 after surgery
  procalcitonin measurement
Systemic clinical evaluation | Day of surgery
  urine excretion rate measurement
Systemic clinical evaluation | Day 7 after surgery
  urine excretion rate measurement
Systemic clinical evaluation | Day 14 after surgery
  urine excretion rate measurement
Histoarchitecture evaluation | Day of surgery
  Haematoxylin & Eosin staining
Histoarchitecture evaluation | Day 14 after surgery
  Haematoxylin & Eosin staining
Histoarchitecture evaluation | Day of surgery
  Movat's Pentachrome staining
Histoarchitecture evaluation | Day 14 after surgery
  Movat's Pentachrome staining
Immunohistochemistry | Day of surgery
  collagen-1 labelling
Immunohistochemistry | Day 14 after surgery
  collagen-1 labelling
Immunohistochemistry | Day of surgery
  collagen-3 labelling
Immunohistochemistry | Day 14 after surgery
  collagen-3 labelling
Immunohistochemistry | Day of surgery
  von Willebrand labelling
Immunohistochemistry | Day 14 after surgery
  von Willebrand labelling
Immunohistochemistry | Day of surgery
  alpha-Smooth Muscle Actin labelling
Immunohistochemistry | Day 14 after surgery
  alpha-Smooth Muscle Actin labelling
Wound healing relative gene expression | Day of surgery
  TGFB1
Wound healing relative gene expression | Day 14 after surgery
  TGFB1
Wound healing relative gene expression | Day of surgery
  TGFB3
Wound healing relative gene expression | Day 14 after surgery
  TGFB3
Wound healing relative gene expression | Day of surgery
  Wnt4
Wound healing relative gene expression | Day 14 after surgery
  Wnt4
Wound healing relative gene expression | Day of surgery
  CTNNB1
Wound healing relative gene expression | Day 14 after surgery
  CTNNB1
Wound healing relative gene expression | Day of surgery
  MMP2
Wound healing relative gene expression | Day 14 after surgery
  MMP2
Wound healing relative gene expression | Day of surgery
  MMP9
Wound healing relative gene expression | Day 14 after surgery
  MMP9

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided